CLINICAL TRIAL: NCT05657925
Title: Randomized, Prospective, Placebo-Controlled, Crossover Study of Ondansetron in the Prevention of Sleep Syncope: The Nineth Prevention of Syncope Trial (POST9)
Brief Title: Study of Ondansetron in the Prevention of Sleep Syncope: The Nineth Prevention of Syncope Trial (POST9)
Acronym: POST9
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: POST9
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Sleep Syncope
Keywords: Ondansetron
MeSH Terms: interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ondansetron (Active Comparator): ondansetron 8 mg prn sublingually when awakening with nausea. as per the FDA label for ondansetron.
  Interventions: Drug: ondansetron 8 mg
- Placebo (Placebo Comparator): Matching placebo will be identical in appearance to the active treatment pill.
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: ondansetron 8 mg — Ondansetron 8 mg prn sublingually when awakening with nausea. as per the FDA label for ondansetron.
  Arms: Ondansetron
Drug: Matching placebo — Matching placebo will be identical in appearance to the active treatment pill
  Arms: Placebo

SUMMARY:
At least 5% of patients with vasovagal syncope also have Sleep Syncope. Patients awake from sleep with profound malaise and gastrointestinal vagal symptoms. About 75% have severe nausea and about 40% have lower abdominal cramps. Some faint while supine, but most find their symptoms so severe that they rise quickly and hurry to the bathroom. Sometime either on the way to the toilet, near it, or shortly afterwards they faint. The nausea is followed by vomiting, and the cramps by watery diarrhea. After relief the patients remain presyncopal, diaphoretic, and tired. Almost all patients also have clinical vasovagal syncope during daytime hours.

The cause of this is unknown. Orthostatic stress cannot be a factor in triggering the event, and in isolated case reports it occurs during non-REM sleep. There is no classic provocative situation of pain, the sight of trauma, or the presence of medical settings. These suggest the importance of central processes and the reduced likelihood that strategies that target maintaining preload (such as with midodrine and fludrocortisone) would be helpful. As well, midodrine is avoided during the night.

Recently the investigators reasoned that if the investigators could rapidly suppress the nausea patients could remain supine, wait out the nausea, and not faint with orthostatic stress. Ondansetron is a potent anti-nausea medication that has rapidly dissolving preparations. Nine patients were instructed to keep one at the bedside, insert it upon waking up with nausea, remain in bed, and raise their legs (if possible). There was partial success with ondansetron 4 mg and complete success with ondansetron 8 mg. This remarkable but anecdotal observation requires formal testing.

Research Objectives: the investigators will test the hypothesis that ondansetron 8 mg prn sublingually on awakening with moderate to severe nausea prevents loss of consciousness in patients with prior Sleep Syncope who awaken with malaise and nausea.

Study Design & Methodology: The main study will be a placebo-controlled, double-blind, randomized, crossover clinical trial. The primary outcome will be the progression of awakening with nausea to syncope. Thirty patients with Sleep Syncope will be randomized 1:1 to receive packages of either ondansetron 8 mg sublingual tablets or matching placebo. They will each receive 3 boxes of 10 tabs, with refills available if needed. Each crossover period will last 6 months.

In a substudy the investigators will test whether the predominant disturbed physiology is bradycardia, decreased venous return, or decreased systemic vascular resistance. This will be assessed using a unique, small, wearable blood pressure sensor that can be rapidly donned on the ear. It records heart rate and beat-to-beat waveforms, which permit estimating stroke volume, systemic vascular resistance, and cardiac output. the investigators will record these variables in all patients continuously from when the device is put on until 30 minutes afterwards. the investigators hypothesize that unlike during syncope provoked by head-up tilt testing, here there will be no decrease in preload until patients arise, and that the main physiologic disturbance during syncope is hypotension due to decreased preload superimposed on heart rate collapse.

Anticipated Outcomes: If successful, this research would be i) the first to report a well-tolerated and highly effective treatment for most sleep syncope, and ii) the first to report the physiology of brain-initiated vasovagal syncope in the community outside a laboratory environment.

DETAILED DESCRIPTION:
Trial interventions: Randomization will be to ondansetron 8 mg sublingual tablets or matching placebo tablets kept at the bedside, to be used upon awakening with premonitory nausea. This is a commonly used dose for rapid treatment of nausea.

Randomization: Patients will be randomized into two treatment groups will be carried out centrally with a randomization scheme using a computerized algorithm. Medication containers will be filled and labelled with the randomization code number centrally. The investigators will complete a screening log of eligible but nonrandomized patients that will contain demographic data and the reason for non-randomization.

Followup: Study nurse coordinators will see the patients in clinic at baseline, 3 months, 6 months, 9 months, and 12 months. The 6-month visit will be the visit during which the patients will be crossed over from one arm to the other. The total study duration will be 52 weeks for each participant. Patients will be asked to notify the study nurse if they experience a premonitory nausea awakening either with or without an ensuing syncope. Pill counts will be conducted to confirm the number of events.

ELIGIBILITY:
Inclusion Criteria:

1. Syncope according to the American College of Cardiology Guidelines 2017
2. ≥1 Sleep Syncope in the year preceding enrolment
3. ≥-2 points on the Calgary Syncope Symptom Score for Structurally Normal Hearts
4. Age ≥ 18 years with informed consent.

Exclusion Criteria:

1. An inability to give informed consent
2. pregnancy,
3. unwilling or unable to use adequate birth control while on study drug
4. QT interval exceeding 500 ms in the absence of correctable factors.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
nausea event causing the patient to awake and prevented from progressing to syncope | Within 12 months period of the study
  One nausea event causing the patient to awake and prevented from progressing to syncope

SECONDARY OUTCOMES:
In a substudy we will test whether the predominant disturbed physiology is bradycardia, decreased venous return, or decreased systemic vascular resistance | Within 12 months period of the study
  This will be assessed using a unique, small wearable blood pressure sensor that can be donned rapidly on the ear.
Hospital Anxiety and Depression Scale (HADS) | every 6 months of the study up to 12 months
  The total score is out of 42, (21 per subscale). Scores are derived by summing responses for each of the two subscales or for the scale as a whole Higher scores indicate greater levels of anxiety or depression. The total HADS score may be regarded as a global measure of psychological distress
Generalized Anxiety Disorder score | every 6 months of the study up to 12 months
  The GAD-7 is useful in primary care and mental health settings as a screening tool and symptom severity measure for the four most common anxiety disorders (Generalized Anxiety Disorder, Panic Disorder, Social Phobia and PostTraumatic Stress Disorder).
  It is 70-90% sensitive and 80-90% specific across disorders / cutoffs (see Evidence section for more).
  Higher GAD-7 scores correlate with disability and functional impairment (in measures such as work productivity and health care utilization)
EQ-5D-3L | every 6 months of the study up to 12 months
  The EQ-5D-3L classification system consists of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression, each with three levels: no problems "1", moderate problems "2", and severe problems "3". Each health state is described as a vector of these five dimensions. With 3 levels for each dimension, the EQ-5D-3L describes 243 distinct health states, with 11111 being the best health state (full health), and 33333 the worst health state.
  In addition to the classification system, each of the instruments also includes a visual analogue scale (EQ VAS). The EQ VAS records the respondent's self-rated health on a visual analogue scale from 0 to 100, whereby 0 indicates 'the worst health you can imagine', and 100 'the best health you can imagine'. This information can be used as a quantitative measure of health as judged by the individual respondents.
Impact of Syncope on Quality of Life | every 6 months of the study up to 12 months
  The ISQL is a brief valid measure of the impact of syncope on quality of life. It measures impairment, fear, depression, and physical limitations, and correlates with recent syncope frequency.
The Short-Form (SF-36) Health Survey | every 6 months of the study up to 12 months
  The SF-36 is a multi-purpose survey designed to capture adult patients' perceptions of their own health and well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No